CLINICAL TRIAL: NCT00877617
Title: Assessment of Quality of Life in Men With High Risk Localized Prostate Cancer Undergoing Neoadjuvant Investigational Therapy
Brief Title: Quality of Life in Men With High Risk Localized Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0305
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: Quality of Life; QOL; Questionnaire; High Risk localized Prostate Cancer; HRLPC; Neoadjuvant Investigational Therapy; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- QOL Questionnaire
  Interventions: Behavioral: QOL Questionnaire

INTERVENTIONS:
Behavioral: QOL Questionnaire — Mailed survey.

SUMMARY:
Primary Objectives:

1. To describe patient quality of life (QOL) related to bladder, bowel, and sexual function, as well as mental and physical health, in patients who received neoadjuvant investigational therapies prior to radical prostatectomy (RP) for high risk clinically localized prostate cancer (HRCLPC).
2. To identify medical and demographic variables that are related with quality of life, e.g., hormonal or non-hormonal neoadjuvant treatment, time since surgery, disease recurrence, subsequent treatment, age, ethnicity, and socioeconomic status.

Secondary Objectives:

1. To describe treatment satisfaction expressed by patients who have received neoadjuvant investigational therapies prior to radical prostatectomy for high risk clinically localized prostate cancer.

DETAILED DESCRIPTION:
Regardless of the survival benefit that a proposed treatment affords a patient, if it results in a poor QOL, it may not be considered a reasonable option. To assess this critical issue, QOL surveys have been developed to determine the post-therapy impact of a given treatment.

In prostate cancer, one of the most widely used validated survey instruments is the Expanded Prostate Cancer Index Composite (EPIC) .8 It contains 4 primary domains that elicit details regarding urinary, bowel, sexual, and hormonal function. The EPIC questionnaire has been widely applied, although it has not been administered to patients undergoing neoadjuvant investigational therapies prior to radical prostatectomy for HRCLPC. Obtaining this information will be important for counseling patients considering similar trials in the future since it will reflect long-term outcomes for functional recovery and mental health-two key concerns of patients deciding whether to enter clinical trials. Furthermore, researchers will be able to stratify these outcomes based on the specific treatment arm to possibly determine how to optimize outcomes while reducing negative impacts of a given therapy.

This is a cross-sectional descriptive study of the QOL of prostatectomy patients who have received neoadjuvant treatment. Anticipated 131 patients will receive a brief survey by to complete and return by mail to M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patient who participated in one of the following neoadjuvant treatment trials:

  * DM96-140 - A Safety Study of TNP-470 Followed by Radical Prostatectomy for Patients with Locally Advanced Adenocarcinoma of the Prostate
  * DM97-095 - A Tolerance & Efficacy Study of Adenoviral Vector Expressing Wild-type P53 (AD-P53) Preoperative Administration Intraprostatically in Patients with Locally Advanced Prostate Cancer Followed by a Radical Prostatectomy
  * ID00-089 - A Tolerance and Efficacy Trial of Preoperative Thalidomide Treatment Followed By Radical Retropubic Prostatectomy (RRP) In Select Patients With Locally Advanced Prostate Cancer
  * ID97-046 - Preoperative Chemotherapy Followed by Radical Prostatectomy for Patients with Locally Advanced Adenocarcinoma of the Prostate
  * ID99-061- A Randomized Trial of Preoperative Chemotherapy and Androgen Ablation Compared to Androgen Ablation Alone Followed by Radical Prostatectomy for Select Patients with Locally Advanced Adenocarcinoma of the Prostate The study will include those patients who completed preoperative therapy and radical prostatectomy.
* Men over the age of 40 years.

Exclusion Criteria:

* Patients that did not undergo both preoperative therapy and a radical prostatectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M.D.Anderson Cancer Center prostate cancer patients who have received neoadjuvant investigational therapies prior to radical prostatectomy for high risk clinically localized prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Quality of life (QOL) variables related to bladder, bowel, and sexual function, as well as mental and physical health, in patients who received neoadjuvant investigational therapies prior to radical prostatectomy (RP) for HRCLPC. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Curtis A. Pettaway, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org